CLINICAL TRIAL: NCT02097134
Title: A Multi-institutional Feasibility Study of Intra-arterial Chemotherapy Given in the Ophthalmic Artery of Children With Retinoblastoma
Brief Title: Intra-arterial Melphalan in Treating Younger Patients With Unilateral Retinoblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARET12P1; NCI-2014-00618 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ARET12P1; ARET12P1 (Other: Children's Oncology Group); ARET12P1 (Other: CTEP); U10CA180886 (NIH); U10CA098543 (NIH)
Record Dates: First submitted 2014-03-25; First posted 2014-03-26 (Estimated); Results first posted 2018-06-26 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Unilateral Retinoblastoma
MeSH Terms: interventions — Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (melphalan) (Experimental): Patients receive melphalan IA on day 1. Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Melphalan

INTERVENTIONS:
Drug: Melphalan — Given IA
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813

SUMMARY:
This pilot clinical trial studies whether unilateral group D retinoblastoma, or retinoblastoma affecting one eye that has spread to the inner jelly like part of the eye, can be treated with a new technique for delivering chemotherapy directly into the blood vessel that supplies the affected eye. This new technique is called intra-arterial injection. Giving melphalan via intra-arterial injection may make it less likely that children will need surgery to remove the eye and may reduce the amount of treatment side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To study the feasibility of delivering melphalan directly into the ophthalmic artery in children with newly diagnosed unilateral group D retinoblastoma, who would otherwise be considered for enucleation.

SECONDARY OBJECTIVES:

I. To estimate the ocular salvage rate after treatment with intra-arterial melphalan in children with newly diagnosed unilateral retinoblastoma with group D disease.

II. To evaluate the toxicities and adverse events associated with delivering multiple doses of intra-arterial chemotherapy.

III. To evaluate vision outcomes in children treated with intra-arterial chemotherapy.

IV. To monitor the rate of the development of metastatic disease while on protocol therapy.

TERTIARY OBJECTIVES:

I. To evaluate the effects of intra-arterial therapy on the histopathology of eyes enucleated for progression.

OUTLINE:

Patients receive melphalan intra-arterially (IA) on day 1. Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 4 months for 1 year, every 6 months for 1 year, and then periodically for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with unilateral group D retinoblastoma
* Magnetic resonance imaging (MRI) (or computed tomography [CT] if MRI is not available) of the brain must be performed within 14 days prior to study entry
* Diagnostic examination under anesthesia (EUA) must be performed within 14 days prior to study entry
* Rapid central review confirmation of group D disease based on RetCam images from diagnostic EUA must be obtained before starting treatment
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2
* Patients must have a life expectancy of >= 8 weeks
* Patients must have adequate renal function, defined as:

  * Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or
  * A serum creatinine based on age/gender as follows:

    * 1 month to < 6 months: 0.4 mg/dL
    * 6 months to < 1 year: 0.5 mg/dL
    * 1 to < 2 years: 0.6 mg/dL
    * 2 to < 6 years: 0.8 mg/dL
    * 6 to < 10 years: 1 mg/dL
    * 10 to < 13 years: 1.2 mg/dL
    * 13 to < 16 years: 1.5 mg/dL (male); 1.4 mg/dL (female)
    * >= 16 years: 1.7 mg/dL (male); 1.4 mg/dL (female)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 2.5 x upper limit of normal (ULN) for age

Exclusion Criteria:

* Patients with bilateral disease
* Unilateral retinoblastoma with group A, B, C, or E eyes
* Prior chemotherapy or radiation therapy for this disease (laser and cryotherapy are allowed and are not considered exclusion criteria)
* Clinical or neuroimaging evidence of extraocular disease or orbital optic nerve involvement

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-10-31 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murali M Chintagumpala, Principal Investigator — Children's Oncology Group
Locations (12):
- United States (12):
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Yale University, New Haven, Connecticut
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Melphalan: Patients receive melphalan intra-arterial (IA) on day 1. Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Melphalan: Given IA
Period: Overall Study
Arm/Group | Melphalan
Started | 14
Completed | 5
Not Completed | 9
Not completed — Physician Decision | 4
Not completed — Non-Protocol Therapy | 1
Not completed — Progressive Disease | 3
Not completed — Refusal of Further Protocol Therapy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Melphalan
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.92 (0.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Experiencing Feasibility Failure
Description: Feasibility failure is defined as a) interventional radiologist is unable to access the ophthalmic artery for the 1st chemotherapy administration for any reason; b) patient develops central retinal artery occlusion after the 1st or 2nd course that does not reopen by the time the next injection is due; or c) the patient cannot receive all three treatments because of Common Terminology Criteria for Adverse Events (CTCAE) complications grade III or IV that are considered possibly, probably or likely related treatment.
Time Frame: Up to 4 months
Population: All Patients who are eligible and evaluable for the feasibility outcome are included in this outcome
Measure: Number; unit: participants
Arm/Group | Melphalan
Number analyzed (Participants) | 12
participants | 4

2. Secondary Outcome: Incidence of Grade 3 or Higher CTCAE Adverse Events Associated With Multiple Doses of IA Chemotherapy
Description: The percentage of patients with at least 1 occurrence of grade 3 or higher CTCAE adverse experience will be provided. Ineligible patients or patients who do not receive any protocol therapy are excluded from reporting of adverse events.
Time Frame: Up to 30 days after completion of study treatment
Population: One patient who did not receive protocol therapy was excluded.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Groups:
- Melphalan: Patients will receive 1 intra-arterial injection (IA) of melphalan every 21- 30 days. Injections may be repeated every 21-30 days (up to a maximum of 3 cycles) assuming the patients meets the criteria to begin the next cycle.
Arm/Group | Melphalan
Number analyzed (Participants) | 13
Percentage of patients | 38 [18 to 64]

3. Secondary Outcome: Probability of Ocular Salvage
Description: A patient will be considered an ocular-salvage success if enucleation because of disease progression or toxicity is not required during the 2 years following enrollment.
Time Frame: 2 years
Population: One patient who did not receive protocol therapy was excluded. Two patients who were lost to follow-up or follow-up was terminated electively prior to 2 years by patient or parent preference were excluded.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Melphalan
Number analyzed (Participants) | 11
Percentage of patients | 36 [15 to 65]

4. Secondary Outcome: Rate of Metastases of Retinoblastoma
Description: The percentage of patients who experience metastases of retinoblastoma will be estimated. Ineligible patients or patients who do not receive any protocol therapy are excluded from this analysis
Time Frame: Up to 2 years
Population: One patient who did not receive protocol therapy was excluded.
Measure: Number; unit: Percentage of Patients
Arm/Group | Melphalan
Number analyzed (Participants) | 13
Percentage of Patients | 0

5. Secondary Outcome: Vision Acuity, Assessed According to the Amblyopia Treatment Study Visual Acuity Testing Protocol
Description: Estimated by the average visual acuity amongst patients evaluated with a 95% confidence interval.
Time Frame: 1 year after therapy
Population: The study was terminated at stage I since the therapy was considered not feasible to deliver.
  No patients had this data available. Patients either had affected eye enucleated, or did not complete protocol therapy.
Arm/Group | Melphalan
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 4 months
Description: The Other Adverse Events field contains Common Terminology Criteria for Adverse Events (CTCAEs) reported on protocol therapy, excluding those that were reported as Serious Adverse Events. The Serious Adverse Events field contains NCI CTCAEs submitted via expedited reporting (NCI AdEERs / CAeRs).
Arm/Group | Melphalan
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 2/14
Other Adverse Events (participants affected / at risk) | 3/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Melphalan (N=14)
Hypotension (Vascular disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Melphalan (N=14)
Anaphylaxis (Immune system disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-30): https://cdn.clinicaltrials.gov/large-docs/34/NCT02097134/Prot_SAP_000.pdf